CLINICAL TRIAL: NCT05141357
Title: A Phase 2 Study to Assess the Safety and Efficacy of HBI-8000 in Combination With Pembrolizumab for Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC)
Brief Title: A Study of HBI-8000 (Tucidinostat) With Pembrolizumab in Non-Small Cell Lung Cancer
Acronym: HBI-8000
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow Recruitment
Sponsor: HUYABIO International, LLC. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HBI-8000-305
Record Dates: First submitted 2021-11-19; First posted 2021-12-02 (Actual); Results first posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Non Small Cell Lung Cancer
Keywords: HBI-8000; Pembrolizumab; NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — HBI-8000; pembrolizumab; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- HBI-8000 in combination with pembrolizumab (Experimental): HBI-8000 - 30 mg/dose, orally twice a week; Pembrolizumab - 400 mg every 6 weeks or 200 mg every 3 weeks according to Prescribing Information and institutional practice
  Interventions: Drug: HBI-8000 in combination with pembrolizumab

INTERVENTIONS:
Drug: HBI-8000 in combination with pembrolizumab — Participants will take 30 mg of HBI-8000 by mouth every 3-4 days on a twice weekly (BIW) schedule. Pembrolizumab will be administered at 400 mg IV every 6 weeks (Q6W) or 200 mg IV every 3 weeks (Q3W) according to Prescribing Information and institution's prescribing practice for pembrolizumab.
  Other Names: tucidinostat; Keytruda®; pembrolizumab

SUMMARY:
A Phase 2 Study to Assess the Safety and Efficacy of HBI-8000 in Combination with Pembrolizumab for Advanced or Metastatic Non-Small Cell Lung Cancer (NSCLC)

DETAILED DESCRIPTION:
This Phase 2 study evaluates HBI-8000, a histone deacetylase inhibitor (HDACi) in combination with pembrolizumab for the treatment of patients with advanced or metastatic non-small cell lung cancer who possess programmed death ligand 1 (PD-L1) expression Tumor Proportion Score (TPS) of 1% or greater.

The Treatment Phase allowed for up to 24 months of treatment (cycles were 21 days), providing the subject did not experience disease progression or unacceptable toxicity.

ELIGIBILITY:
Inclusion Criteria

1. Adults at least 18 years of age.
2. Eastern Cooperative Oncology Group (ECOG) performance status ≤2.
3. Histopathologically confirmed diagnosis of NSCLC PD-L1 expression TPS ≥1% as determined by an FDA-approved test.
4. Have at least one measurable target lesion as defined by RECIST v.1.1.
5. Have not received immune checkpoint inhibitor therapy or more than one regimen of chemotherapy for advanced or metastatic disease. Subjects who have previously received immune checkpoint inhibitor therapy in the adjuvant or neoadjuvant setting may be allowed if disease progression occurred >6 months after the last dose and no clinically significant immune related toxicities leading to treatment discontinuation were observed.
6. Prior adjuvant or neoadjuvant systemic therapy with chemotherapy, EGFR or ALK mutation directed therapy must have been completed >4 weeks before Cycle 1 Day 1 (C1D1) dosing and recovered from all treatment related toxicity.
7. Any prior palliative radiotherapy or minor surgery must be completed at least 2 weeks and 1 week respectively before C1D1 dosing and recovered from all treatment related toxicities.
8. Adequate major organ functions at baseline as evidenced by laboratory findings within 14 days prior to C1D1 study drug administration as defined below:

   1. White blood cells (WBC) ≥3000/μL, neutrophils ≥1500/μL, platelets ≥100×103/μL, hemoglobin ≥9.0 g/dL, independent of transfusion.
   2. Serum creatinine ≤1.5 mg/dL, normal electrolytes, phosphorus, and calcium.
   3. Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤3 × upper limit of normal (ULN), alkaline phosphatase ≤2.5 × ULN unless bone metastases present, bilirubin ≤1.5 × ULN (unless known Gilbert's disease where it must be ≤3 × ULN) and serum albumin ≥3.0 g/dL.
   4. Thyroid stimulating hormone (TSH) within normal limits.
9. Life expectancy ≥12 weeks.
10. A negative serum pregnancy test at baseline for women of childbearing potential (WOCBP).
11. Women of childbearing potential. (WOCBP), non-surgically sterile or premenopausal female capable of becoming pregnant and men (due to potential risk of drug exposure through the ejaculate) must agree to use an acceptable method of contraception while enrolled on this study, and for a period of 5 months following the last dose of treatment. Acceptable methods of birth control in this trial include 2 highly effective methods of birth control (as determined by the Investigator; one of the methods must be a barrier technique) or abstinence.
12. Have the ability to understand and the willingness to sign a written informed consent document.

Exclusion Criteria

1. History of Grade ≥3 hypersensitivity reactions to monoclonal antibodies.
2. History of a cardiovascular illness including: QT interval corrected by heart rate using Fridericia's correction formula (QTcF) >450 ms in male or >470 ms in female, congenital long QT syndrome, congestive heart failure (New York Heart Association Grade III or IV) (Protocol Appendix 2); unstable angina or myocardial infarction within the previous 6 months; or symptomatic cardiac arrhythmia despite medical management.
3. Uncontrolled hypertension, systolic blood pressure (SBP) >160 mmHg or diastolic blood pressure (DBP) >100 mmHg.
4. Central nervous system metastasis or leptomeningeal disease except when treatment for brain metastasis is completed >14 days prior to C1D1 and stable for ≥4 weeks on <10 mg daily prednisone or equivalent.
5. History of hemorrhagic diarrhea, inflammatory bowel disease, active uncontrolled peptic ulcer disease or bowel resection that affects absorption of orally administered drugs.
6. Recurrent pleural effusion requiring repetitive palliative thoracentesis within 3 months prior to study entry, except for subjects with a pleurex port.
7. Active, known, or suspected autoimmune disease, or history of immune-mediated toxicity leading to treatment discontinuation, except for type I diabetes mellitus, hypothyroidism only requiring hormone replacement or skin disorders (such as vitiligo, psoriasis, or alopecia) not requiring systemic therapy.
8. Active pneumonitis, history of non-infectious pneumonitis that required treatment with steroids, or history of interstitial lung disease.
9. Active uncontrolled bacterial, viral, or fungal infection requiring systemic therapy.
10. Known history of testing positive for human immunodeficiency virus (HIV), known acquired immunodeficiency syndrome (AIDS).
11. Active hepatitis B (hepatitis B surface antigen [HBVsAg] positive), or hepatitis C (HCV antibody test or serum hepatitis C ribonucleic acid [RNA] positive).
12. Received approved live vaccines within 30 days of planned C1D1. Inactivated viral vaccines or vaccines based on subviral component are allowed; however intranasal influenza vaccines (e.g., Flu-Mist) are not allowed. COVID-19 vaccination should be administered >7 days before C1D1.
13. Any condition requiring chronic systemic treatment with either corticosteroids (>10 mg daily prednisone equivalents) or other immunosuppressive medications, or steroids use within 14 days of study drug administration. Inhaled or topical steroids are permitted.
14. Use of other investigational agent (drug not marketed for any indication) within 28 days or at least 5 half-lives (whichever is shorter) before study drug administration.
15. Pregnant or breast-feeding women.
16. Second malignancy unless in remission for 2 years; subjects with non-melanomatous skin cancer, carcinoma in situ of the cervix treated with curative intent, or curatively treated prostate cancer with prostate-specific antigen (PSA) <2.0 ng/mL can be included.
17. Underlying medical conditions that, in the Investigator's opinion, will make the administration of study drug hazardous or obscure the interpretation of toxicity determination or adverse events.
18. Unwilling or unable to comply with procedures required in this protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2022-02-15 (Actual); Primary Completion 2023-04-19 (Actual); Study Completion 2023-04-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gloria Lee, MD, PhD, Study Director — HUYABIO International, LLC.
Locations (7):
- United States (7):
  - Western Regional Medical Center, Goodyear, Arizona
  - CBCC Global Research, Inc at Comprehensive Blood and Cancer Center, Bakersfield, California
  - Hematology Oncology Associates Of The Treasure Coast, Port Saint Lucie, Florida
  - Southeastern Regional Medical Center, Newnan, Georgia
  - Midewestern Regional Medical Center, LLC, Zion, Illinois
  - Cotton O'Neil Clinical Research Center, Topeka, Kansas
  - Frederick Health-JMSCI, Frederick, Maryland

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a multicenter (9 sites in the US: hospital, regional medical, and research centers), open label, Phase 2 study of HBI 8000 in combination with an approved dose of pembrolizumab as a first line checkpoint inhibitor therapy for advanced or metastatic non-small cell lung cancer (NSCLC). Recruitment was from 15Feb 2022 to 01Sep2022. In December 2022, enrollment was suspended.
Pre-assignment Details: Subjects had to satisfy screening criteria prior to treatment with HBI-8000 + Pembrolizumab. The screening period could be up to 28 days and was comprised of assessing medical history, concomitant therapies, clinical laboratory testing, and other clinical assessments to document the subject met all inclusion criteria and none of the exclusion criteria.
Groups:
- HBI-8000 in Combination With Pembrolizumab: HBI-8000 in combination with pembrolizumab: Participants will take 30 mg of HBI-8000 by mouth every 3-4 days on a twice weekly (BIW) schedule. Pembrolizumab was administered at 400 mg IV every 6 weeks (Q6W) or 200 mg IV every 3 weeks (Q3W) according to Prescribing Information and institution's prescribing practice for pembrolizumab.
Period: Overall Study
Arm/Group | HBI-8000 in Combination With Pembrolizumab
Started | 5
Completed | 0
Not Completed | 5
Not completed — Adverse Event | 3
Not completed — Lack of Efficacy | 2

BASELINE CHARACTERISTICS:
Arm/Group | HBI-8000 in Combination With Pembrolizumab
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 0
  >=65 years | 5
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 4
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 4
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: Safety and Tolerability of HBI-8000 When Administered in Combination With Standard Dose and Regimen of Pembrolizumab
Description: Number of participants experiencing treatment-emergent adverse events (TEAEs) graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0
Time Frame: From the start of treatment until 30 days after the last dose of HBI-8000, up to approximately 13 months
Measure: Count of Participants; unit: Participants
Arm/Group | HBI-8000 in Combination With Pembrolizumab
Number analyzed (Participants) | 5
Participants
  Subjects experiencing TEAEs | 5
  Subjects not experiencing TEAEs | 0

ADVERSE EVENTS:
Time Frame: Up to approximately 13 months
Arm/Group | HBI-8000 in Combination With Pembrolizumab
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 3/5
Other Adverse Events (participants affected / at risk) | 5/5
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HBI-8000 in Combination With Pembrolizumab (N=5)
Diarrhoea (Gastrointestinal disorders) | 1
Gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
COVID-19 pneumonia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Hypotension (Vascular disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | HBI-8000 in Combination With Pembrolizumab (N=5)
Anaemia (Blood and lymphatic system disorders) | 3
Iron deficiency anemia (Blood and lymphatic system disorders) | 3
Thrombocytopenia (Blood and lymphatic system disorders) | 3
Atrial fibrillation (Cardiac disorders) | 1
Cardiac failure (Cardiac disorders) | 1
Pericardial effusion (Cardiac disorders) | 1
Sinus tachycardia (Cardiac disorders) | 2
Tachycardia (Cardiac disorders) | 1
Ear pain (Ear and labyrinth disorders) | 1
Middle ear effusion (Ear and labyrinth disorders) | 1
Hypothyroidism (Endocrine disorders) | 1
Periorbital pain (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Abdominal distension (Gastrointestinal disorders) | 1
Anal incontinence (Gastrointestinal disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 4
Feces discolored (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Lip pain (Gastrointestinal disorders) | 1
Lower gastrointestinal haemorrhage (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Oral lichen planus (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 2
Asthenia (General disorders) | 1
Fatigue (General disorders) | 2
Non-cardiac chest pain (General disorders) | 1
Oedema peripheral (General disorders) | 2
Pyrexia (General disorders) | 1
COVID-19 pneumonia (Infections and infestations) | 1
Cellulitis (Infections and infestations) | 1
Fungal skin infection (Infections and infestations) | 1
Otitis media (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 2
Sinusitis (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Fall (Injury, poisoning and procedural complications) | 1
Amylase increased (Investigations) | 2
Eastern Cooperative Oncology Group performance status worsened (Investigations) | 1
Lipase increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 1
Platelet count decreased (Investigations) | 2
Weight decreased (Investigations) | 2
White blood cell count decreased (Investigations) | 2
White blood cells urine positive (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 4
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hypophosphataemia (Metabolism and nutrition disorders) | 1
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Squamous cell carcinoma of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Dizziness (Nervous system disorders) | 2
Nerve compression (Nervous system disorders) | 1
Insomnia (Psychiatric disorders) | 1
Haematuria (Renal and urinary disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 1
Wheezing (Respiratory, thoracic and mediastinal disorders) | 1
Lichen planus (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2
Urticaria (Skin and subcutaneous tissue disorders) | 1
Hypotension (Vascular disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-27): https://cdn.clinicaltrials.gov/large-docs/57/NCT05141357/Prot_SAP_000.pdf